CLINICAL TRIAL: NCT06065358
Title: Ovarian Tumor Organotypic Slices Cultures for functionAl Drug Testing and Therapy Response Prediction
Acronym: TOSCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4128
Record Dates: First submitted 2023-06-21; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional, prospective, monocentric (Experimental)
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor biopsy — Patients with advanced suspected HGSOC will be considered eligible (FIGO stage from III C or greater). At the time of surgery, patients' disease extension will be assessed with the Fagotti score (PIV) and the Vizzielli score (VS). Only patients who are not considered operable in the first place, will be enrolled. Samples will be taken during surgery that will take place in the operating rooms of oncological gynaecology.

SUMMARY:
Ex vivo organotypic tumor slice cultures (OTSC) have unique characteristics in terms of tissue processing time and the maintenance of original microenvironment. Moreover, drug screening has been successfully performed on OTSC in a clinically meaningful time window.

For these reasons, we designed a study to assess the feasibility of establishing OTSC in OC patients and the concordance between ex vivo sensitivity and in vivo treatment response. If proven effective and reliable, OTSC could be introduced into clinical practice as empirical predictor of patients' response to platinum.

DETAILED DESCRIPTION:
Most patients with ovarian cancer (OC) present with advanced stage and severe symptoms. The standard of care is based on an association between surgery and platinum-based chemotherapy, to which targeted therapies have been added since 2014. Despite significantly improved outcomes, there are still 15-20% of patients resistant to platinum-based chemotherapy without many therapeutic options and poor prognosis. It is urgent to select this population thus limiting useless undesirable effects and exploring more effective therapeutic options before clinical conditions worsen. To date, there are no validated predictive markers of primary platinum refractory or resistant disease and traditional cancer models are currently incompatible with treatment time window in this clinical setting.

Among cancer models, ex vivo organotypic tumor slice cultures (OTSC) have unique characteristics in terms of tissue processing time and the maintenance of original microenvironment. Moreover, drug screening has been successfully performed on OTSC in a clinically meaningful time window.

For these reasons, we designed a study to assess the feasibility of establishing OTSC in OC patients and the concordance between ex vivo sensitivity and in vivo treatment response. If proven effective and reliable, OTSC could be introduced into clinical practice as empirical predictor of patients' response to platinum.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative clinical, serological and radiologic suspicion of International Federation of Gynecology and Obstetrics (FIGO) stage IIIC or greater ovarian, fallopian tube, or primary peritoneal cancer;
2. Age over 18 years;
3. Estimated life expectancy of at least 4 weeks;
4. Fagotti score (PIV) > 8 or patients not considered operable in the first place for any reasons;
5. Histologic diagnoses of epithelial ovarian cancer at frozen section.

Exclusion Criteria:

1. Non- epithelial histology at frozen section;
2. Patients enrolled in other clinical trials.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
To test the effect of chemotherapeutic drugs on ovarian cancer cell cultures. | 24 months
  To evaluate the concordance of chemotherapy drug response in ovarian cancer patients treated in vivo and in cell culture of tumor tissue harvested and treated in vitro.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No